CLINICAL TRIAL: NCT02125487
Title: The Use of Hybrid Simulation (HS) of the Breast in Teaching Clinical Breast Examination (CBE) to Medical Students.
Brief Title: Hybrid Simulation in Teaching Clinical Breast Examination
Acronym: HS-CBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Rana Sharara, Simulation Program Director, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: PED.RS1.03
Record Dates: First submitted 2014-03-18; First posted 2014-04-29 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Medical Education; Clinical Breast Examination; Medical Simulation; Standardized Patient
Keywords: Clinical Breast Examination; Breast Cancer detection; Breast Simulator; Hybrid Simulation; Patient Simulation; Standardized Patient; Medical student education; Health Communication; Communication Barriers; Cultural competency; Cultural; Middle East; Lebanon

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-Fidelity Simulation (Active Comparator): Teaching using traditional method
  Interventions: Behavioral: Teaching using traditional method
- Hybrid Simulation (Experimental): Teaching using Hybrid Simulation of breast examination
  Interventions: Behavioral: Teaching using Hybrid Simulation of breast examination

INTERVENTIONS:
Behavioral: Teaching using Hybrid Simulation of breast examination — Students in the "intervention/experimental" group will receive the regular lecture given at the American University of Beirut and will attend a screening of an educational video on the technique of CBE, in addition to the hybrid simulation teaching activities in the simulation lab (standardized patient wearing breast examination simulator jackets)
  Other Names: Standardized Patient wearing breast jacket
  Arms: Hybrid Simulation
Behavioral: Teaching using traditional method — Students in the "control" group will receive the regular lecture given at the American University of Beirut and will attend the usual simulation lab teaching activities (single breast silicone model without any actors). The only new introduction to the curriculum is an educational video on the technique of CBE.
  Other Names: Lecture with low-fidelity breast model
  Arms: Low-Fidelity Simulation

SUMMARY:
The purpose of this study is to determine whether the use of hybrid simulation of the breast are more effective in teaching CBE technique and culturally sensitive doctor-patient communication skills to medical students than the traditional method.

DETAILED DESCRIPTION:
Breast cancer is a Lebanese national problem. Campaigns for mammography screening are effective but recommendations on breast examinations screening for breast tumors are lacking. On one hand, the Lebanese population is culturally diverse, with women's beliefs ranging from liberal to extremely conservative. On the other hand, Clinical Breast Examination (CBE) is traditionally taught to medicine III students in a lecture, followed by practice on a low-fidelity breast model. The opportunity to clinically practice CBE depends on patient availability and her willingness to be examined by students. This is further limited by some Lebanese women's cultural and religious beliefs. Little is known about the effect of patient cultural practices on the efficacy of CBE.

In this project, we focus on the need for an effective educational tool for teaching CBE to physicians-in-training. The proposed teaching method in this study is hybrid simulation: breast model jacket (simulator) worn by a trained actress (standardized patient, SP). In this study, we compare this standardized educational tool to the traditional teaching method which consists of a lecture and training on a low-fidelity (unrealistic) breast model on a desk (no SP).

We hypothesize that the use of this hybrid simulation tool, as compared to the traditional teaching method, will result in a more complete CBE, better lesion detection and improved culturally sensitive communication skills in terms of awareness of, and ability to deal with, cultural differences related to breast examination.

In order to do so, we will evaluate medical students' performance and examine their attitudes and cultural competencies when they perform CBEs on 3 culturally different standardized patients using hybrid simulation scenarios. Through an experimental design that minimizes biases related to selection of students (randomized controlled), we will compare hybrid simulation (intervention) with low-fidelity simulation (control) in teaching CBE.

Medicine-III students rotating in the Obstetrics and Gynecology department at the American University of Beirut Medical Center (AUBMC) will be asked to participate; they are free to refuse without any effect on their grades in the rotation. The students will be assessed in an Objective Structured Clinical Examination (OSCE) setting similar to their usual oral clinical exams but not contributory to their academic evaluation in the Faculty of Medicine. The OSCE setting will include encounters with 3 culturally different Standardized Patients (1 "outgoing" woman, 1 with "chador", and 1 moderately conservative woman). The assessment tools are questionnaires that are either objective (filled by SP) or self-reporting (filled by students) about (1) met learning objectives, (2) student's attitude, and (3) clinical cultural competency.

ELIGIBILITY:
Inclusion Criteria:

* Third year medical students (Med III) at the American University of Beirut
* Rotating in the Obstetrics and Gynecology department at the American University of Beirut Medical Center

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
CBE completeness (in OSCE) | Each participant will be assessed once, after an average of 2-3 weeks following the intervention (teaching activity)
  SPs will be objectively grading the students on a scoring sheet

SECONDARY OUTCOMES:
Student's attitude about the teaching activity | Each participant will be assessed once, after an average of 2-3 weeks following the intervention (teaching activity)
  Self-reported questionnaires
Cultural communication skills (in OSCE) | Each participant will be assessed once, after an average of 2-3 weeks following the intervention (teaching activity)
  SPs will be objectively grading the students on a scoring sheet
Student's attitude about the assessment activity (OSCE) | On the day of the assessment activity, after an average of 2-3 weeks following the intervention (teaching activity)
  Self-reported questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Karim Sleiman, MD, Study Director — American University of Beirut Medical Center; Rana Sharara-Chami, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

REFERENCES:
- [Background] Coleman EA, Stewart CB, Wilson S, Cantrell MJ, O'Sullivan P, Carthron DO, Wood LC. An evaluation of standardized patients in improving clinical breast examinations for military women. Cancer Nurs. 2004 Nov-Dec;27(6):474-82. doi: 10.1097/00002820-200411000-00007. PMID 15640625
- [Background] Costanza ME, Luckmann R, Quirk ME, Clemow L, White MJ, Stoddard AM. The effectiveness of using standardized patients to improve community physician skills in mammography counseling and clinical breast exam. Prev Med. 1999 Oct;29(4):241-8. doi: 10.1006/pmed.1999.0544. PMID 10547049
- [Background] Facione NC, Katapodi M. Culture as an influence on breast cancer screening and early detection. Semin Oncol Nurs. 2000 Aug;16(3):238-47. doi: 10.1053/sonc.2000.8118. PMID 10967796
- [Background] Pugh CM, Salud LH; Association for Surgical Education. Fear of missing a lesion: use of simulated breast models to decrease student anxiety when learning clinical breast examinations. Am J Surg. 2007 Jun;193(6):766-70. doi: 10.1016/j.amjsurg.2006.12.033. PMID 17512293
- [Background] Schubart JR, Erdahl L, Smith JS Jr, Purichia H, Kauffman GL, Kass RB. Use of breast simulators compared with standardized patients in teaching the clinical breast examination to medical students. J Surg Educ. 2012 May-Jun;69(3):416-22. doi: 10.1016/j.jsurg.2011.10.005. Epub 2011 Nov 25. PMID 22483147
- [Derived] Nassif J, Sleiman AK, Nassar AH, Naamani S, Sharara-Chami R. Hybrid Simulation in Teaching Clinical Breast Examination to Medical Students. J Cancer Educ. 2019 Feb;34(1):194-200. doi: 10.1007/s13187-017-1287-3. PMID 29019167